CLINICAL TRIAL: NCT00396812
Title: An Open Label, Single Arm, Single Center, Phase I/II Trial of Rituximab (a Monoclonal Antibody to CD20) for the Treatment of Early Rheumatoid Arthritis
Brief Title: Rituximab for the Treatment of Early Rheumatoid Arthritis (RA)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The perceived risk-benefit ratio for individuals with early active RA
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ARA04
Record Dates: First submitted 2006-11-06; First posted 2006-11-08 (Estimated); Results first posted 2012-11-14 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Autoimmune disease; Biologic response modifiers; Disease-modifying antirheumatic drugs (DMARDS); Immune system; Rheumatoid arthritis (RA); Rituximab (anti-CD20 monoclonal antibodies)
MeSH Terms: conditions — Arthritis, Rheumatoid; Autoimmune Diseases | interventions — Rituximab

ARMS (1):
- Rituximab (Experimental)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Participants to receive an intravenous infusion of rituximab (1 gram ) fourteen days apart, at baseline (Day 0) and at Week 2.
  Concomitant treatments to be administered at a dose and frequency prescribed per protocol include methotrexate (MTX) and folic or folinic acid.
  Other Names: Anti-CD20 antibody therapy; Rituxan

SUMMARY:
Rheumatoid arthritis (RA) is a chronic inflammatory disease characterized by joint swelling, pain, stiffness, damage, and ultimately loss of joint function. Scientists estimate that about 1.3 million people (0.6 percent) of the U.S. adult population have RA. Current therapies target the immune system early in the disease process before joint damage occurs, and include drugs such as methotrexate (MTX) and tumor necrosis factor (TNF)-blocking agents. Rituximab is a disease-modifying antirheumatic drug (DMARD) recently approved by the FDA for use in combination with MTX for treatment of moderately to severely active RA in patients who have had an inadequate response to TNF-blocking agents, in an effort to try to slow the course of the disease. This study will examine the effects of rituximab on the immune response and disease activity in participants with early RA who have not been treated with any disease-modifying agent. In addition, the safety and tolerability of rituximab in this population will be examined.

DETAILED DESCRIPTION:
RA is an inflammatory disease that causes pain, swelling, stiffness, and loss of function in the joints. It occurs when the immune system, which normally defends the body from invading organisms, turns its attack against the membrane lining the joints. RA is commonly managed by DMARDs initiated early in the disease process, before irreversible joint damage occurs. The most common DMARD prescribed in the United States is MTX; this drug is well tolerated and has better efficacy compared to other DMARDs, but is inadequate in providing lasting improvement in individuals with RA. In patients with an inadequate response to MTX alone, the use of biologic agents, including TNF-blocking agents in combination with MTX, has become a standard therapeutic approach.

Rituximab (anti-CD20) is a man-made antibody used to treat certain types of cancer. The drug blocks the CD20 antigen found on the surface of B cells and is known to deplete B cells when administered intravenously. Previous research suggests B-cell activity is important in pathogenesis of RA, so B-cell depletion may decrease inflammation and other symptoms of RA. Rituximab has recently been approved by the FDA for use in combination with MTX for treatment of patients with moderately to severely active RA who have had an inadequate response to TNF-blocking agents. This study will examine the effects of rituximab on the immune response and disease activity in patients with early active RA who have not been treated with any disease-modifying agent. Levels of B and T cells and other markers of disease activity will be monitored during the study. The safety and tolerability of rituximab in this DMARD-naive population will be examined.

The expected duration of this study is 2.5 years. All participants will receive two intravenous infusions of rituximab in an outpatient setting at study entry and Week 2. Throughout the study, participants will receive MTX, systemic corticosteroids, and folic or folinic acid. MTX dosing will be re-evaluated by disease activity scores every month until Month 6 and again at Months 8, 10, and 12. Systemic corticosteroid doses will be modified based on the participant's health while in the study. Use of nonsteroidal anti-inflammatory drugs (NSAIDs) is permitted, but NSAID doses should not be changed during the study, if at all possible. NSAIDs will not be provided by this study.

There will be a maximum of 2 screening visits before study treatment, a baseline visit (Day 0), and 11 study visits. A physical exam, assessment for adverse events, and blood collection will occur at all study visits. Kidney and liver function tests and rheumatologic evaluations will occur at most study visits; participants will also be asked to complete a questionnaire on their health at most study visits. Arthroscopy (knee biopsy) on the more inflamed knee will occur at baseline and Month 3. Participants will be contacted by telephone the day after each arthroscopy and rituximab infusion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA, as defined by fulfilling at least four of seven American College of Rheumatology (ACR) criteria
* Positive for rheumatoid factor (RF) and/or anticyclic citrullinated peptide (CCP)
* The presence of arthritis symptoms for more than 6 weeks but less than 1 year
* Active RA, as defined by at least four swollen joints, at least four tender joints, and either an erythrocyte sedimentation rate (ESR) of greater than 30 mm/hr OR C-reactive protein level greater than 1.0 mg/dL (normal less than 0.4)
* Willing to adhere to the study requirements
* Willing to use acceptable effective forms of contraception

Exclusion Criteria:

* Allergy to methotrexate (MTX)
* Previous exposure to anti-CD20 monoclonal antibody (mAb) or other type(s) of mAb therapy
* Previous disease-modifying anti-rheumatic drugs (DMARD) therapy
* Previous use of a biologic agent
* Currently taking daily oral steroid doses of greater than 7.5 milligrams (mg)
* Receipt of intra-articular injections within 4 weeks prior to study entry
* Current peptic ulcer disease (PUD)
* Unwilling to stop drinking alcohol (ETOH)
* History of alcohol or substance abuse
* Active infection, or chronic or persistent infection that might worsen with immunosuppressive treatment (e.g., Human Immunodeficiency Virus [HIV], hepatitis B virus [HBV], hepatitis C virus [HCV], tuberculosis [TB])
* Interstitial lung disease observed by chest x-ray [chest radiograph]
* Known coronary artery disease or significant cardiac arrhythmias or severe congestive heart failure (New York Heart Association [NYHA] classes III or IV)
* Definitive diagnosis of another autoimmune rheumatologic disease (e.g., systemic lupus erythematosus [SLE], scleroderma, primary Sjögren's syndrome, primary vasculitis)
* History of immunoglobulin E (IgE)-mediated or non-IgE-mediated hypersensitivity or known anaphylaxis to mouse proteins
* History of cancer. Exception: participants with previous resected basal or squamous cell carcinoma, treated cervical dysplasia, or treated in situ Grade I cervical cancer within 5 years prior to study entry are not excluded from study eligibility
* History of positive purified protein derivative (PPD) test (i.e., positive tuberculosis [TB] test) without treatment for TB infection or chemoprophylaxis for TB exposure
* History of inflamed pancreas
* Live vaccine within 3 months of study entry
* Certain abnormal laboratory values
* Require certain medications
* Any psychiatric disorder that would prevent a participant from providing informed consent
* Any condition or treatment (including biologic therapies) that, in the opinion of the investigator, may place the participant at unacceptable risk during the study
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Striebich, MD, PhD, Study Chair — Rheumatology Division, University of Colorado Health Sciences Center; Robert D. D'Ambrosia, MD, Principal Investigator — Department of Orthopedics, University of Colorado Health Sciences Center
Locations (1):
- University of Colorado Health Sciences Center, Denver, Colorado, United States

REFERENCES:
- [Background] De Vita S, Quartuccio L. Treatment of rheumatoid arthritis with rituximab: an update and possible indications. Autoimmun Rev. 2006 Aug;5(7):443-8. doi: 10.1016/j.autrev.2006.02.007. Epub 2006 Mar 15. PMID 16920570
- [Background] Eisenberg R, Albert D. B-cell targeted therapies in rheumatoid arthritis and systemic lupus erythematosus. Nat Clin Pract Rheumatol. 2006 Jan;2(1):20-7. doi: 10.1038/ncprheum0042. PMID 16932648
- [Background] Isenberg DA. B cell targeted therapies in autoimmune diseases. J Rheumatol Suppl. 2006 May;77:24-8. PMID 16652442
- [Background] Looney RJ. B cell-targeted therapy for rheumatoid arthritis: an update on the evidence. Drugs. 2006;66(5):625-39. doi: 10.2165/00003495-200666050-00004. PMID 16620141

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 subjects were to be enrolled into the open label early Rheumatoid Arthritis trial at one site in the US. Enrollment occurred in 2008 but the study was terminated early due to Genentech's announcement regarding rituximab's risk-benefit ratio for individuals with early active Rheumatoid Arthritis.
Period: Overall Study
Arm/Group | Rituximab
Started | 4
Completed | 3 (4 subjects completed treatment, but 1 subject terminated early due to disease progression)
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43.3 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 4
Disease Activity Score 28 -Erythrocyte Sedimentation Rate (DAS28-ESR) [Mean (Standard Deviation); unit: Score on a scale] — The DAS28-ESR is a score on a scale (0 to 10) measure of the subject's disease activity. It is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity (mm), and ESR (mm/hour). Flares in disease activity are defined as an increase greater than 1.2 in this score and remission is defined as achieving a DAS28-ESR score of less than 2.6
  Score on a scale | 5.1 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Disease Activity Score- Erythrocyte Sedimentation Rate (DAS28-ESR) at Week 48
Description: The DAS28-ESR is a score on a scale (0 to 10) that is a measure of the subject's disease activity. It is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity (mm), and ESR (mm/hour). Lower score indicates less disease activity. Flares in disease activity are defined as an increase in this score of greater than 1.2 and remission is defined as achieving a DAS28-ESR score of less than 2.6.
Time Frame: Baseline (Day 0), Week 48
Population: All subjects who receive at least one dose of study treatment and attended Day 0 and Week 48 visits
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 3
Score on a scale | -1.5 (1.5)

2. Primary Outcome: Change From Baseline in Tender Joint Count Score at Week 48
Description: Tender Joint Count (TJC) is calculated based on tenderness response of 28 joints. TJC possible values range from 0 to 28. A lower TJC indicates less joint tenderness. Change from baseline is computed as Week 48 value minus baseline value. A negative value in change from baseline indicates an improvement.
Time Frame: Baseline (Day 0), Week 48
Population: All subjects who receive at least one dose of study treatment and attended Day 0 and Week 48 visits
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 3
Units on a scale | 1.3 (8.4)

3. Primary Outcome: Change From Baseline in Swollen Joint Count at Week 48
Description: Swollen Joint Count (SJC) is calculated based on swelling response of 28 joints. SJC possible values range from 0 to 28. A lower SJC indicates less joint swelling. Change from baseline is computed as Week 48 value minus baseline value. A negative value in change from baseline indicates an improvement.
Time Frame: Baseline (Day 0), Week 48
Population: All subjects who receive at least one dose of study treatment and attended Day 0 and Week 48 visits
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 3
Units on a scale | -4.7 (1.2)

4. Primary Outcome: Change From Baseline in Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS) at Week 48
Description: Change from Baseline in PAAP-VAS (0 to 100 millimeters visual analog scale, 0 being no pain and 100 being most severe pain) is computed as the value at Week 48 minus the Baseline value. A negative value in change from Baseline indicates an improvement.
Time Frame: Baseline (Day 0), Week 48
Population: All subjects who receive at least one dose of study treatment and attended Day 0 and Week 48 visits
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rituximab
Number analyzed (Participants) | 3
mm | -2.3 (4.7)

5. Primary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity- Visual Analog Scale (PtGADA-VAS) at Week 48
Description: Change from Baseline in PtGADA-VAS (0 to 100 millimeters visual analog scale, 0 being no symptoms and 100 being severe symptoms) is computed as the value at Week 48 minus the Baseline value. A negative value in change from Baseline indicates an improvement.
Time Frame: Baseline (Day 0), Week 48
Population: All subjects who receive at least one dose of study treatment and attended Day 0 and Week 48 visits
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rituximab
Number analyzed (Participants) | 3
mm | -1.2 (4.6)

6. Primary Outcome: Change From Baseline in Physician's Global Assessment of Patient's Disease Activity- Visual Analog Scale (PhGADA-VAS) at Week 48
Description: Change from Baseline in PhGADA-VAS (0 to 100 millimeters visual analog scale, 0 being no symptoms and 100 being severe symptoms) is computed as the value at Week 48 minus the Baseline value. A negative value in change from Baseline indicates an improvement.
Time Frame: Baseline (Day 0), Week 48
Population: All subjects who receive at least one dose of study treatment and attended Day 0 and Week 48 visits
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rituximab
Number analyzed (Participants) | 3
mm | -2.4 (1.7)

7. Primary Outcome: Change From Baseline in the Short Form 36 (SF-36) Physical and Mental Health Component Summary Scores (PCS and MCS) at Week 48
Description: SF-36 measures health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores: PCS=physical functioning, role-physical, bodily pain, and general health; MCS=vitality, social functioning, role-emotional, and mental health. Scoring is done for both subscores and summary scores. For both, 0=worst score (or quality of life) and 100=best score. Change from baseline is computed as the value at Week 48 minus the baseline value. A positive value in change from Baseline indicates an improvement and a negative value worsening.
Time Frame: Baseline (Day 0), Week 48
Population: All subjects who receive at least one dose of study treatment and attended Day 0 and Week 48 visits
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 3
Units on a scale
  Change in Short-Form-36 Physical Health Score | 14.5 (4.3)
  Change in Short-Form-36 Mental Health Score | -1.2 (12.8)

8. Primary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 48
Description: HAQ-DI is derived based on the mean of individual scores in 8 categories of daily living activities (using 20 questions). Each question is scored 0-3 (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do). In addition, category scores are modified if an aid or device is used, for example, a walker or wheelchair, or help is received from another person in the daily living activities. If an aid or device is used or help is received then a category score of 0 or 1 increases to a category score of 2. A category score of 3 remains a 3 regardless of aids, devices, or help. Scores from each of the 8 categories are totaled. The total score can range from 0 to 24. Change from baseline is computed as the total score at Week 48 minus the baseline total score. A negative value in change from baseline indicates an improvement.
Time Frame: Baseline (Day 0), Week 48
Population: All subjects who receive at least one dose of study treatment and attended Day 0 and Week 48 visits
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 3
Units on a scale | -0.9 (0.3)

9. Primary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Week 48
Description: ESR is a blood test used to monitor therapy in inflammatory diseases such as rheumatoid arthritis and reflects acute phase reactant levels. Active disease in RA is defined by an ESR greater than 30 mm/hr. Change from baseline is computed as the value at Week 48 minus the baseline value. A negative value in change from baseline indicates an improvement.
Time Frame: Baseline (Day 0), Week 48
Population: All subjects who receive at least one dose of study treatment and attended Day 0 and Week 48 visits
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Rituximab
Number analyzed (Participants) | 3
mm/hr | -24.7 (15.9)

ADVERSE EVENTS:
Time Frame: From the start of steroid taper, when applicable, and otherwise, from 1.)time of the 1st invasive screening procedure (knee arthroscopy) until participant study completion (Wk 48) or 2.)30 days after a participant prematurely withdraws from the study.
Description: This study graded the severity of adverse events experienced by the study participant according to criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 3.0 (June 10, 2003).
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=4)
Tachycardia (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Infusion related reaction (General disorders) | 2 (2)
Parvovirus infection (Infections and infestations) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial terminated early due to rituximab's risk-benefit ratio for individuals with early active Rheumatoid Arthritis. Mechanistic samples were not processed and corresponding endpoints were not assessed. Only descriptive statistics are presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No